CLINICAL TRIAL: NCT00926120
Title: A Phase II, Open-label, Efficacy and Safety Study to Evaluate the Effects of Mogroside Sweetener "PureLo" on Viral Load in Treatment Naïve, Genotype 1 Subjects With Chronic Hepatitis C
Brief Title: The Effects of Mogroside Sweetener on Viral Load in TreatmenT Naive Genotype 1 (GT 1) Subjects CHC
Acronym: PureLo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Stephen A Harrison, Principal Investigator, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.2008.193
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mogroside sweetener (Experimental): All subjects will received Mogroside. Mogroside sweetener administered at a dosage level of 5 g every 6 hours for 14 days.
  Interventions: Dietary Supplement: Mogroside sweetener (PureLo)

INTERVENTIONS:
Dietary Supplement: Mogroside sweetener (PureLo) — Mogroside sweetener administered at a dosage level of 5g every 6 hours for 14 days
  Other Names: Pure Lo

SUMMARY:
The purpose of this study is to determine if administering Mogroside Sweetener "PureLo" (the study substance) for 14 days will lower the hepatitis C viral load and liver function alanine aminotransferase (ALT) levels.

DETAILED DESCRIPTION:
The primary objectives of the study are to assess the safety and efficacy of administering Mogroside Sweetener "PureLo" to genotype 1 subjects at a dose level of 5 grams every 6 hours for 14 days on hepatitis C viral load and serum ALT levels. Percentage change in HCV load over the first 48 hours and daily for 14 days and change in serum ALT levels over the two week period of study, will be calculated for each patient. The number of subjects who show a decline in viral load of at least 50% will then be calculated, as will the number of subjects who decrease their serum ALT levels by at least 50%. All efficacy and safety analysis will be conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Serologic evidence of HVC infection by an anti-HCV antibody test.
* Serum HCV RNA quantifiable > 20,000 copies/mL at screening period and demonstrate abnormal ALT > 40 for 6 months.
* No clinical suspicion or radiological evidence of hepatocellular carcinoma and a serum AFP < 50 ng/mL.
* Negative urine pregnancy test for women of childbearing potential documented within the 24-hour period prior to the first dose for test drug.

Exclusion Criteria:

* Interferon with or without RBV therapy at any previous time or any other systemic antiviral therapy or investigational drug > 3 months prior to the first dose of study drug.
* Subjects who are expected to need systemic antiviral therapy at any time during the study are also excluded.
* Positive test at screening for anti-HAV 1gM Ab, HbsAg, anti-HBc IgM Ab, or anti-HIV Ab.
* Documented serum concentrations of ceruloplasmin or Alpha 1-antitrypsin consistent with an increased risk of metabolic liver disease.
* History or other evidence of a medical condition associated with chronic liver disease (e.g., haemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures).
* Women with ongoing pregnancy or breast feeding
* Neutrophil count < 1000 cells/mm3, Hgb <11 g/dL in women or 12 g/dL in men, or platelet count < 80,000 cells/mm3.
* Serum creatinine level > 2 times the upper limit of normal at screening.
* Evidence of alcohol and/or drug abuse within one year of entry.
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquillizer at therapeutic doses for major depression or psychosis, respectively, for at least 4 months at any previous time or any history of the following:

  * a suicidal attempt
  * hospitalization for psychiatric disease, OR
  * a period of disability due to a psychiatric disease.
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematous, autoimmune hemolytic anemia, scleroderma, severe psoriasis, sarcoidosis, etc.).
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease including ascites or hepatic encephalopathy.
* History or other evidence of chronic pulmonary disease associated with functional limitation.
* History of severe cardiac disease.
* History of a severe seizure disorder or current anticonvulsant use.
* Evidence of an active or suspected cancer or a past history of malignancy other than skin cancer.
* History of having received any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤ 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* History of major organ transplantation with an existing functional graft.
* History of thyroid disease poorly controlled on prescribed medications.
* History or other evidence of severe retinopathy.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of administering Mogroside sweetener "PureLo" at a dosage level of 5 g every 6 hours over 15 in subjects with chronic hepatitis C (CHC) with respect to the following: hepatitis C viral load; serum ALT levels. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Harrison, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States